CLINICAL TRIAL: NCT07026864
Title: Project #1: MRI-guided Bladder Cancer Preservation Program
Brief Title: MRI-Guided Bladder Preservation Program For Patients With Muscle Invasive Bladder Cancer
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Clinica Universidad de Navarra, Universidad de Navarra (Other)
Responsible Party: Principal Investigator, Rafael Martínez Monge, Scientific Director, Radiation Oncology Department, Clinica Universidad de Navarra, Universidad de Navarra
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024.110
Record Dates: First submitted 2025-06-10; First posted 2025-06-18 (Actual); Last update posted 2025-08-24 (Actual); Status verified 2025-06

CONDITIONS: Muscle Invasive Bladder Cancer (MIBC)
Keywords: Muscle Invasive Bladder Cancer; Bladder Preservation; Radiation Therapy; MR-Guided Radiation Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MRI-guided Bladder Cancer Preservation Program (Experimental)
  Interventions: Radiation: MR-guided Radiation Therapy

INTERVENTIONS:
Radiation: MR-guided Radiation Therapy — MR-guided Radiation Therapy

SUMMARY:
The goal of this clinical trial is to learn if the use of MRI-guided irradiation increases the rates of bladder preservation as well as to decrease complications in patients with muscle invasive bladder cancer who wish to retain their bladders

DETAILED DESCRIPTION:
HYPOTHESIS The implementation of Magnetic Resonance Image Guided Radiotherapy (MRgRT) into a Bladder Preservation Program maximizes treatment objectives rates due to the better visualization and online dose-adaptation of the TURBT cavity.

Rationale In the radiation setting, MRI provides superior soft tissue contrast compared to standard onboard X-ray imaging improving inter- and intra- observer delineation variation (Noel et al., 2015). MRgRT offers the opportunity to adapt the plan at each fraction to the anatomical changes seen (Henke et al., 2018). This is especially important in bladder tumors where bladder is subject to large interfractional position changes as well as intrafractional shape and size variation since the on-board median filling rate is close to 2 ml/min. This requires that intrafraction bladder filling has to be successfully accommodated in order to maintain adequate target coverage (Dees-Ribbers et al., 2014). It is hypothesized therefore that MRgRT facilitates tumor boost and partial bladder irradiation approaches (Hafeez et al., 2016; Vestergaard et al., 2016).

MRgRT has been shown to be feasible. Authors reported that the full online adaptive planning workflow based on the anatomy seen at each fraction was delivered within 45 min. Intra-fraction bladder filling did not compromise target coverage. Patients reported acceptable tolerance of treatment (Hunt et al., 2020).

Primary Objectives A. To achieve pathological complete response rate in 95% of the patients. B. To decrease urinary grade 3 or greater toxicity below 3% and rectal grade 3 or greater toxicity below 1%.

Secondary Objectives A. Determination of blood and urine biomarkers of treatment response and toxicity .

B. Determination of radiomics biomarkers of treatment response and toxicity . C. Determination of urinary functionality with IPSS and Bladder Control Self-Assessment Questionnaire

ELIGIBILITY:
Inclusion Criteria:

1. Patients with T2-T3N0M0 unifocal bladder cancer of any histologic subtype except squamous cell carcinoma or adenocarcinoma (Janopaul-Naylor et al., 2021) treated the maximal TURBT and able to tolerate concurrent chemoradiotherapy. Selected patients with high risk of common iliac involvement (T4 disease and/or limited N+ disease and/or LVSI+ status) able to receive the following treatment may be included as well. Additional criteria include:
2. Karnofsky performance status > 70 with medical condition not contraindicating treatment with radical intent including maximal TURBT and concomitant chemotherapy;
3. WBC equal or greater than 3500 mm3; platelet count equal or greater than 135000 mm3; hemoglobin equal or greater than 10 gr/L; BUN equal or less than 20; serum creatinine equal or less than 2.0.

Exclusion Criteria:

1. Prior radiation therapy to the target areas;
2. Inability to undergo a MRI exam

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2030-07-01 (Estimated); Study Completion 2030-07-01 (Estimated)

PRIMARY OUTCOMES:
Pathological complete response rate and Urinary and Rectal Toxicity | Five years
  A. To achieve pathological complete response rate in 95% of the patients. B. To decrease urinary grade 3 or greater toxicity below 3% and rectal grade 3 or greater toxicity below 1%.

SECONDARY OUTCOMES:
Blood and urine biomarkers, Radiomics biomarkers and PROMs | 5 years
  A. Determination of blood and urine biomarkers of treatment response and toxicity .
  B. Determination of radiomics biomarkers of treatment response and toxicity . C. Determination of urinary functionality with IPSS and Bladder Control Self-Assessment Questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Rafael Martínez-Monge, M.D., Principal Investigator — Clínica Universidad de Navarra; Marta Moreno-Jiménez, M.D., Principal Investigator — Clínica Universidad de Navarra

IPD SHARING:
Plan to Share IPD: Yes
On request
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: July 1st, 2025 - June 30th, 2030
Access Criteria: On request